CLINICAL TRIAL: NCT01557647
Title: Inhaled Treprostinil for the Treatment of Pulmonary Arterial Hypertension: A Phase III, International, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Event-Driven Study to Evaluate the Safety and Efficacy of Inhaled Treprostinil.
Brief Title: Safety and Efficacy of Inhaled Treprostinil in Patients With PAH
Acronym: INTREPID
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIN-PH-302
Record Dates: First submitted 2012-03-14; First posted 2012-03-19 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inhaled treprostinil (Experimental)
  Interventions: Drug: Inhaled treprostinil
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled treprostinil — 0.6mg/mL treprostinil for inhalation solution. Titrated up to 12 breaths QID.
  Arms: inhaled treprostinil
Drug: Placebo — placebo inhalation solution
  Arms: placebo

SUMMARY:
To evaluate the effect of inhaled treprostinil compared to placebo on exercise capacity and time to clinical worsening.

ELIGIBILITY:
Eligible subjects must:

* Be between 18 and 75 years of age at Screening (as defined by date of informed consent is signed),
* Have a diagnosis of idiopathic or heritable PAH, PAH associated with connective tissue disease (CTD), PAH associated with repaired congenital systemic-to-pulmonary shunts (at least 1 year since repair) or human immunodeficiency virus (HIV) infection, or PAH associated with appetite suppressant or toxin use.
* Be treatment naïve, or receiving background PAH therapies (e.g., phosphodiesterase type-5 inhibitor (PDE-5i)and / or endothelin receptor antagonist (ERA)) for less than 1 year prior to Screening.
* Have a 6MWD at Baseline (as measured by the mean value of two 6MWT separated by at least 24 hours, but no more than 14 days) that is between 150 - 500 meters, inclusive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | 6 months

SECONDARY OUTCOMES:
Time to clinical worsening | 1 day to 2.5 years.